CLINICAL TRIAL: NCT04252664
Title: A Phase 3 Randomized, Double-blind, Placebo-controlled Multicenter Study to Evaluate the Efficacy and Safety of Remdesivir in Hospitalized Adult Patients With Mild and Moderate COVID-19.
Brief Title: A Trial of Remdesivir in Adults With Mild and Moderate COVID-19
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: The epidemic of COVID-19 has been controlled well at present, no eligible patients can be recruitted.
Sponsor: Capital Medical University (Other)
Collaborators: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Bin Cao, Professor, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAP-China remdesivir 1
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: COVID-19; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — remdesivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remdesivir group (Experimental): active remdesivir
  Interventions: Drug: Remdesivir
- Control group (Placebo Comparator): Placebos matched remdesivir
  Interventions: Drug: Remdesivir placebo

INTERVENTIONS:
Drug: Remdesivir — RDV 200 mg loading dose on day 1 is given, followed by 100 mg iv once-daily maintenance doses for 9 days.
  Other Names: GS-5734
  Arms: Remdesivir group
Drug: Remdesivir placebo — RDV placebo 200 mg loading dose on day 1 is given, followed by 100 mg iv once-daily maintenance doses for 9 days.
  Arms: Control group

SUMMARY:
In December 2019, Wuhan, in Hubei province, China, became the center of an outbreak of pneumonia of unknown cause. In a short time, Chinese scientists had shared the genome information of a novel coronavirus (SARS-CoV-2) from these pneumonia patients and developed a real-time reverse transcription PCR (real-time RT-PCR) diagnostic assay.

Given no specific antiviral therapy for COVID-19 and the availability of remdesvir as a potential antiviral agent based on pre-clinical studies in SARS-CoV and MERS-CoV infections, this randomized, controlled, double blind trial will evaluate the efficacy and safety of remdesivir in patients hospitalized with mild or moderate COVID-19.

DETAILED DESCRIPTION:
In December 2019, Wuhan, in Hubei province, China, became the center of an outbreak of pneumonia of unknown cause. In a short time, Chinese scientists had shared the genome information of a novel coronavirus (SARS-CoV-2) from these pneumonia patients and developed a real-time reverse transcription PCR (real time RT-PCR) diagnostic assay.

Whilst the outbreak is likely to have started from a zoonotic transmission event associated with a large seafood market that also traded in live wild animals, it soon became clear that person-to-person transmission was also occurring. The number of cases of COVID-19 identified in Wuhan increased markedly over the later part of January 2020, with cases identified in multiple other Provinces of China and internationally. Mathematical models of the expansion phase of the epidemic suggested that sustained person-to-person transmission is occurring, and the R-zero is substantially above 1, the level required for a self-sustaining epidemic in human populations.

The clinical spectrum of COVID-19 appears to be wide, encompassing asymptomatic infection, a mild upper respiratory tract illness, and severe viral pneumonia with respiratory failure and even death. Although the per infection risk of severe disease remains to be determined, and may differ from the initial reports of 10-15%, the large number of cases in Wuhan has resulted in a large number of patients hospitalised with pneumonia. Progression from prodromal symptoms (usually fever, fatigue, cough) to severe pneumonia requiring supplementary oxygen support, mechanical ventilation, or in some cases ECMO appears to occur most commonly during the second week of illness in association with persistent viral RNA detection. This provides a window of opportunity to test candidate antiviral therapeutics.

This new coronavirus, and previous experiences with SARS and MERS-CoV, highlight the need for therapeutics for human coronavirus infections that can improve clinical outcomes, reduce risk of disease progression, speed recovery, and reduce the requirements for intensive supportive care and prolonged hospitalisation. In addition, treatments for mild cases to reduce the duration of illness and infectivity may also be of value were COVID-19 to become pandemic and/or endemic in human populations.

Given no specific antiviral therapy for COVID-19 and the availability of remdesvir as a potential antiviral agent based on pre-clinical studies in SARS-CoV and MERS-CoV infections, this randomized, controlled, double blind trial will evaluate the efficacy and safety of remdesivir in patients hospitalized with mild or moderate COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at time of signing Informed Consent Form
2. Laboratory (RT-PCR) confirmed COVID-19.
3. Lung involvement confirmed with chest imaging
4. Hospitalised with:

   * Fever - ≥36.7℃ -axilla or Oral temperature ≥ 38.0 ℃ or ≥38.6°C tympanic or rectal or
   * And at least one of Respiratory rate >24/min Or Cough
5. ≤8 days since illness onset
6. Willingness of study participant to accept randomization to any assigned treatment arm.
7. Must agree not to enroll in another study of an investigational agent prior to completion of Day 28 of study.

Exclusion Criteria:

1. Physician makes a decision that trial involvement is not in patients' best interest, or any condition that does not allow the protocol to be followed safely.
2. Severe liver disease (e.g. Child Pugh score ≥ C, AST>5 times upper limit)
3. SaO2/SPO2≤94% in room air condition, or the Pa02/Fi02 ratio <300mgHg
4. Known allergic reaction to remdesivir
5. Patients with known severe renal impairment (estimated glomerular filtration rate ≤30 mL/min/1.73 m2) or receiving continuous renal replacement therapy, hemodialysis, peritoneal dialysis
6. Pregnant or breastfeeding, or positive pregnancy test in a predose examination
7. Will be transferred to another hospital which is not the study site within 72 hours.
8. Receipt of any experimental treatment for COVID-19 within the 30 days prior to the time of the screening evaluation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2020-02-12 (Actual); Primary Completion 2020-04-10 (Estimated); Study Completion 2020-04-27 (Estimated)

PRIMARY OUTCOMES:
Time to Clinical recoveryTime to Clinical Recovery (TTCR) | up to 28 days
  TTCR is defined as the time (in hours) from initiation of study treatment (active or placebo) until normalisation of fever, respiratory rate, and oxygen saturation, and alleviation of cough, sustained for at least 72 hours, or live hospital discharge, whichever comes first.
  Normalisation and alleviation criteria:
  * Fever - <37°C,
  * Respiratory rate - ≤24/minute on room air,
  * Oxygen saturation - >94% on room air,
  * Cough - mild or absent on a patient reported scale of severe, moderate, mild, absent.

SECONDARY OUTCOMES:
All cause mortality | up to 28 days
  baseline SpO2 during screening, PaO2/FiO2 <300mmHg or a respiratory rate ≥ 24 breaths per min without supplemental oxygen
Frequency of respiratory progression | up to 28 days
  Defined as SPO2≤ 94% on room air or PaO2/FiO2 <300mmHg and requirement for supplemental oxygen or more advanced ventilator support.
Time to defervescence (in those with fever at enrolment) | up to 28 days
Time to cough reported as mild or absent (in those with cough at enrolment rated severe or moderate) | up to 28 days
Time to dyspnea reported as mild or absent (on a scale of severe, moderate, mild absent, in those with dyspnoea at enrolment rated as severe or moderate,) | up to 28 days
Frequency of requirement for supplemental oxygen or non-invasive ventilation | up to 28 days
Time to 2019-nCoV RT-PCR negative in upper respiratory tract specimen | up to 28 days
Change (reduction) in 2019-nCoV viral load in upper respiratory tract specimen as assessed by area under viral load curve. | up to 28 days
Frequency of requirement for mechanical ventilation | up to 28 days
Frequency of serious adverse events | up to 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Jin Yin-tan hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Grundeis F, Ansems K, Dahms K, Thieme V, Metzendorf MI, Skoetz N, Benstoem C, Mikolajewska A, Griesel M, Fichtner F, Stegemann M. Remdesivir for the treatment of COVID-19. Cochrane Database Syst Rev. 2023 Jan 25;1(1):CD014962. doi: 10.1002/14651858.CD014962.pub2. PMID 36695483
- [Derived] Ansems K, Grundeis F, Dahms K, Mikolajewska A, Thieme V, Piechotta V, Metzendorf MI, Stegemann M, Benstoem C, Fichtner F. Remdesivir for the treatment of COVID-19. Cochrane Database Syst Rev. 2021 Aug 5;8(8):CD014962. doi: 10.1002/14651858.CD014962. PMID 34350582